CLINICAL TRIAL: NCT04273204
Title: Does One-Leg-Standing Duration Have a Relationship With Gross Motor Function Measurement Scores and Stance Phase for Unilateral Spastic Children
Brief Title: Relationships Between OLST, GMFM and Pedobarographic Values in CP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Kültür University (Other)
Collaborators: Istanbul University (Other)
Responsible Party: Principal Investigator, Gamze Ertürk, Research assistant, Istanbul Kültür University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2017/397
Record Dates: First submitted 2020-02-11; First posted 2020-02-18 (Actual); Last update posted 2020-02-18 (Actual); Status verified 2020-02

CONDITIONS: Cerebral Palsy
Keywords: cerebral palsy,; gait,; Gross Motor Function Measurement,; stability,; foot pressure
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- UCP Group (Experimental)
  Interventions: Diagnostic Test: one leg standing test, gross motor function measurement, pedobarographic measurement
- Control Group (Other)
  Interventions: Diagnostic Test: one leg standing test, gross motor function measurement, pedobarographic measurement

INTERVENTIONS:
Diagnostic Test: one leg standing test, gross motor function measurement, pedobarographic measurement — OLST:During the OLST,the participants were asked to shoes off,place both hands on their hips and look at a point on the wall at eye level.A recording stopwatch was used to assess their standing duration on one leg while keeping the other leg in 90 degrees of knee flexion.The test was stopped when the contralateral foot touched the ground or when the participant broke 90 degrees of knee flexion.The OLST was repeated three times for each leg.GMFM:To assess standing and walking,running and jumping functions of the UCP group,the D and E dimensions of GMFM were utilized by a certificated physiotherapist.Each item was tested by three trials and the best trial was used.Pedobarography:The participants' plantar pressure was analyzed using pedobarography.For each participant, the pedobarography was calibrated before the assessment.During the pedobarographic analysis, the participants walked barefoot in 90 BPM cadence. Three steps were analyzed for each side.

SUMMARY:
The primary aim of this study was to investigate the relationship between the One Leg-Standing Test (OLST) and the Gross Motor Function Measurement (GMFM) and stance phase stability during gait in Unilateral Cerebral Palsy (UCP). The secondary aim was to explore a new well-defined pedobarographic parameter as a functional factor in the stability of stance in gait.

The investigator's hypotheses are (1) OLST has relationship between T2-T1 in children with UCP; (2) OLST has relationship between GMFM D and E.

Eighteen children with UCP and ten typically developing children (TDC) participated in the study. All participants and their legal guardians signed an informed consent form before participating. Firstly, to asses the stability in stance all participants were analyzed by using pedobarographic analysis and the OLST. After analysis, only the UCP group was evaluated with the GMFM. The TDC group was used for comparison of pedobarographic stance phase stability (T2-T1) and OLST values.

ELIGIBILITY:
Inclusion Criteria (for experimental group):

* diagnosed unilateral cerebral palsy
* be able to stand on the affected leg for 0 to 30 seconds

Exclusion Criteria:

* Children with UCP who had Botulinum Toxin-A injections to the lower limbs in the previous six months
* Lower limb surgeries
* Mental disorders

Ages: 7 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 28 (Actual)
Dates: Start 2018-01-10 (Actual); Primary Completion 2018-03-15 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
One leg standing test (OLST) | 1 time, baseline of the study
  During the OLST, the participants were asked to shoes off, place both hands on their hips and look at a point on the wall at eye level. A recording stopwatch was used to assess their standing duration on one leg while keeping the other leg in 90 degrees of knee flexion. The test was stopped when the contralateral foot touched the ground or when the participant broke 90 degrees of knee flexion. The OLST was repeated three times for each leg and the best score was chosen.
Gross Motor Function Measurement (GMFM) | 1 time, baseline of the study
  The Gross Motor Function Measure (GMFM) is an assessment tool designed and evaluated to measure changes in gross motor function over time or with intervention in children with cerebral palsy. Items span the spectrum of gross motor activities in five dimensions.
  A: Lying and Rolling,
  B: Sitting,
  C: Crawling and Kneeling,
  D: Standing, and
  E: Walking, Running and Jumping. In our study, To assess standing and walking, running and jumping functions of the UCP group (GMFCs level I and II), the D and E dimensions of GMFM were utilized by a certificated physiotherapist. Each item was tested by three trials and the best trial was scoring between 0-3 points.
Pedobarographic Measurement | 1 time, baseline of the study
  The participants' plantar pressure was analyzed using pedobarography (Tekscan Inc. Mass. USA) with rectangular shape plates (43.59 x 36.88 x 5.77 cm) and 2288 resistive pressure sensors. For each participant, the pedobarography was calibrated before the assessment. During the pedobarographic analysis, the participants walked barefoot in 90 BPM cadence with the aid of a metronome. Before the pedobarographic analysis, each participant walked three minutes to adapt to the metronome.Three steps were analyzed for each side (affected and unaffected sides) to evaluate the following parameters i) time of peak force in early stance phase (T1), ii) time of peak force of late stance phase (T2), iii) stance phase stability (T2-T1), iv) duration of total stance phase (TS) and v) ratio (T2-T1/TS). A mean value of each parameter was used for statistical analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Kültür University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No